CLINICAL TRIAL: NCT07038915
Title: STRIVE: A Single-arm Phase 2 Study on Treatment of Lung Squamous Cell Carcinoma by Tiragolumab Plus Ivonescimab for Patients Who Progressed on Platinum Doublets and Anti-PD-1/PD-L1
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: 0 participants
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0406; NCI-2025-04492 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Lung Squamous Cell Carcinoma; Anti-PD1/PDL1 Antibody
MeSH Terms: interventions — Tiragolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental): Treatment with Tiragolumab + Ivonescimab
  Interventions: Drug: Tiragolumab; Drug: Ivonescimab

INTERVENTIONS:
Drug: Tiragolumab — Given by IV
Drug: Ivonescimab — Given by IV

SUMMARY:
To learn if the drug combination of tiragolumab and ivonescimab can help to control LSCC that got worse after standard treatment with platinum doublets and anti-PD-1/PD-L1 therapy.

DETAILED DESCRIPTION:
Primary Objectives To determine the objective response rate (ORR) of metastatic LSCC patients who progressed on platinum doublets and anti-PD1/PD-L1 treated with Tiragolumab/Ivonescimab.

Secondary Objectives To evaluate the investigator assessed progression-free survival (PFS) and overall survival (OS) based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 of tiragolumab in combination with ivonescimab To evaluate the duration of response (DoR) of tiragolumab in combination with ivonescimab, as assessed by investigator, based on RECIST v1.1 To evaluate the safety and tolerability of tiragolumab in combination with ivonescimab

ELIGIBILITY:
Eligibility Criteria

1. Voluntarily sign a written informed consent form
2. Age ≥ 18 years old at the time of enrollment
3. Ability of comply with the study protocol, in the investigator's judgement
4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2
5. Expected life expectancy ≥ 3 months
6. Metastatic (Stage IV) NSCLC, according to American Joint Committee on Cancer (AJCC) 8th edition
7. Histologically or cytologically confirmed lung squamous cell carcinoma (LSCC). Participants with mixed histology (eg, adenosquamous) are allowed if there is squamous component.
8. Disease progression during or following treatment with platinum doublets and anti-PD(L)1 containing therapy for metastatic LSCC.
9. At least one measurable noncerebral lesion according to RECIST 1.1. Target lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions since radiotherapy. Sites of biopsy cannot be included as target lesions unless no other measurable lesions are present.
10. Adequate hematologic and end-organ function, defined by the following laboratory test results, obtained within 14 days prior to initiation of study treatment:

    a. Hematology (no blood transfusions or growth factor therapy used within 7 days of the screening CBC): i. Absolute neutrophil count (ANC) ≥ 1.5 × 109/L ii. Platelet count ≥ 100 × 109/L iii. Hemoglobin ≥ 9.0 g/dL iv. Lymphocyte count ≥ 0.5 × 109/L b. Kidneys: i. Creatinine clearance (CrCl) ≥ 50 mL/min using the Cockcroft-Gault formula or estimated glomerular filtration rate (eGFR) value ≥50 mL/min using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation ii. Urine protein < 2+ or 24 hour urine protein quantification < 1.0 g iii. Serum albumin ≥ 25 g/L (2.5 g/dL). c. Liver: i. Serum total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN); For patients with liver metastases or confirmed/suspected Gilbert syndrome: TBIL ≤3 × ULN ii. Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) ≤ 2.5 × ULN; For Participants with liver metastases: AST and ALT ≤ 5 × ULN; For Participants with liver and bone metastases: ALP ≤ 5 ×ULN d. Coagulation: i. For Participants not receiving therapeutic anticoagulation: prothrombin time (PT) or international normalized ratio (INR) ≤ 1.5 x ULN, and partial prothrombin time (PTT) or activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN (unless abnormalities are unrelated to coagulopathy, or prophylactic coagulation) ii. For Participants receiving therapeutic anticoagulation: stable anticoagulant regimen defined as clinical stability on unchanged dose of therapeutic anticoagulation for ≥14 days
11. Negative HIV test at screening with the following exception: individuals with a positive HIV test at screening are eligible provided they are stable on anti-retroviral therapy, have a CD4+ T cell count ≥ 200/uL, and have an undetectable viral load
12. Negative hepatitis B surface antigen (HBsAg) test at screening
13. Positive hepatitis B surface antibody (HBsAb) test at screening, or negative HBsAb at screening accompanied by either of the following:

    1. Negative total hepatitis B core antibody (HBcAb)
    2. Positive total HBcAb test followed by quantitative hepatitis B virus (HBV) DNA < 500 IU/mL The HBV DNA test will be performed only for Participants who have a negative HBsAg test, a negative HBsAb test, and a positive total HBcAb test
14. Negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV RNA test at screening The HCV RNA test will be performed only for Participants who have a positive HCV antibody test
15. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods, and agreement to refrain from donating eggs, as defined below:

    1. Women must remain abstinent or use contraceptive methods with a failure rate of < 1% per year during the treatment period and for 6 months after the final dose of study treatment.

       Women must refrain from donating eggs during this same period.
    2. A woman is considered to be of childbearing potential if she is postmenarchal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause) and has not undergone surgical sterilization (removal of ovaries and/or uterus). The definition of childbearing potential may be adapted for alignment with local guidelines or requirements.
    3. Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.
    4. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post-ovulation methods) and withdrawal are not adequate methods of contraception.
16. For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm, as defined below:

    1. With a female partner of childbearing potential who is not pregnant, men who are not surgically sterile must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period and for 120 days after the final dose of tiragolumab and ivonescimab. Men must refrain from donating sperm during this same period.
    2. With a pregnant female partner, men must remain abstinent or use a condom during the treatment period and for 120 days after the final dose of tiragolumab and ivonescimab to void potential exposure to the embryo.
    3. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post-ovulation methods) and withdrawal are not adequate methods of contraception

Exclusion Criteria

1. Prior treatment with anti-TIGIT antibody therapy
2. Symptomatic central nervous system (CNS) metastases
3. History of leptomeningeal disease
4. Uncontrolled tumor-related pain Participants requiring pain medication must be on a stable regimen at study entry.

   Symptomatic lesions (e.g., bone metastases or metastases causing nerve impingement) amenable to palliative radiotherapy should be treated prior to enrollment. Participants should be recovered from the effects of radiation. There is no required minimum recovery period.

   Asymptomatic metastatic lesions that would likely cause functional deficits or intractable pain with further growth (e.g., epidural metastasis that is not currently associated with spinal cord compression) should be considered for loco-regional therapy if appropriate prior to enrollment.
5. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently) Participants with indwelling catheters (e.g., PleurX) are allowed.
6. Uncontrolled or symptomatic hypercalcemia (ionized calcium >1.5 mmol/L, calcium >12 mg/dL or corrected serum calcium > ULN
7. Active or history of clinically significant autoimmune disease that, in the opinion of the investigator, could compromise the health and safety of the patient if treated with investigational therapy. Notable exceptions include:

   1. Participants with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone
   2. Participants with controlled type 1 diabetes mellitus who are on an insulin regimen
   3. Active or history of adrenal insufficiency on stable steroid regimen
   4. Participants with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only are eligible for the study provided all of following conditions are met:

   i. Disease is well controlled at baseline and requires only low-potency topical corticosteroids ii. No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency oral corticosteroids within the previous 12 months
8. History of bleeding tendencies or coagulopathy and/or clinically significant bleeding symptoms or risk within 4 weeks prior to enrollment, including but not limited to:

   1. Gastrointestinal bleeding
   2. Hemoptysis (defined as coughing up ≥ 1 teaspoon of fresh blood or blood clots) Note: transient hemoptysis associated with diagnostic bronchoscopy is allowed.
   3. Nasal bleeding /epistaxis (bloody nasal discharge is allowed)
   4. Need for therapeutic anticoagulant therapy within 14 days prior to enrollment Note: Prophylactic anticoagulation for DVT/PE or to maintain venous patency is allowed.
   5. Other intermediate to high bleeding risks determined by treating physicians
9. Imaging during the screening period shows that the patient has:

   1. Radiologically documented evidence of major blood vessel invasion or encasement by cancer
   2. Radiographic evidence of intratumor cavitation
10. Active idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted
11. Known active tuberculosis
12. Major surgical procedures or serious trauma within 4 weeks prior to enrollment, or plans for major surgical procedures within 4 weeks after the first dose (as determined by the investigator). Minor local procedures (excluding central venous catheterization and port implantation) within 3 days prior to enrollment
13. Active malignancy other than NSCLC that requires treatment, with the exception of malignancies with a negligible risk of metastasis or death as assessed and confirmed by the study principal investigator (PI). Possible examples include: adequately treated carcinoma in situ of the cervix, non melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or stage I uterine cancer
14. Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment Participants receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
15. Severe infection within 2 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection (including coronavirus disease 2019 [COVID-19]), bacteremia, or severe pneumonia
16. Prior allogeneic stem cell or solid organ transplantation
17. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, in the view of the investigator, contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications
18. Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during study treatment or within 5 months after the final dose of study treatment of tiragolumab or ivonescimab
19. Positive Epstein-Barr virus (EBV) viral capsid antigen immunoglobulin M (IgM) test at screening An EBV polymerase chain reaction (PCR) test should be performed as clinically indicated to screen for acute infection or suspected chronic active infection. Participants with a positive EBV PCR test are excluded.
20. Treatment with investigational therapy within 21 days prior to initiation of study treatment
21. Prior immune-related adverse event resulting in permanent discontinuation of immune checkpoint blockade therapy including but not limited to anti-PD-1, anti-PD-L1 and anti-CTLA4 therapeutic antibodies that, in the view of the investigator, could compromise health and safety of prospective patient if enrolled in the study
22. Inadequately controlled hypertension (defined as systolic blood pressure ≥ 150 mmHg and/or diastolic blood pressure ≥ 100 mmHg). Anti-hypertensive therapy to achieve these parameters is allowable
23. Prior history of hypertensive crisis or hypertensive encephalopathy
24. History of major diseases before enrollment, specifically:

    1. Unstable angina, myocardial infarction, congestive heart failure (New York Heart Association [NYHA] classification ≥ grade 2) or vascular disease (eg, aortic aneurysm at risk of rupture) that required hospitalization within 12 months prior to enrollment, or other cardiac impairment that may affect the safety evaluation of the study drug (eg, poorly controlled arrhythmias, myocardial ischemia)
    2. History of esophageal gastric varices, severe ulcers, wounds that do not heal, abdominal fistula, intra-abdominal abscesses, or acute gastrointestinal bleeding within 6 months before enrollment
    3. History of arterial thromboembolic event, venous thromboembolic event of Grade 3 and above as specified in National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) 5.0, transient ischemic attack, cerebrovascular accident, hypertensive crisis, or hypertensive encephalopathy within 6 months prior to enrollment
    4. Acute exacerbation of chronic obstructive pulmonary disease within 4 weeks before enrollment
    5. History of perforation of the gastrointestinal tract and/or fistula, history of gastrointestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), extensive bowel resection (partial colectomy or extensive small bowel resection) within 6 months prior to enrollment
25. History of intracranial bleeding within 1 year if initiation of treatment
26. Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, < 7 days prior to the first dose of study treatment
27. Serious, non-healing or dehiscing wound, active ulcer, or untreated bone fracture
28. Proteinuria, as demonstrated by urine dipstick or > 1.0 g of protein in a 24-hour urine collection. All Participants with >= 2+ protein on dipstick urinalysis at baseline must undergo a 24-hour urine collection for protein
29. Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and IL-2) within 4 weeks or 5 drug-elimination half-lives (whichever is longer) prior to initiation of study treatment
30. Treatment with systemic immunosuppressive medication (including, but not limited to: corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-alpha agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions: a. Participants who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study after PI confirmation has been obtained b. Participants who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study
31. History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins • Known hypersensitivity to Chinese hamster ovary cell products or to any component of the tiragolumab and ivonescimab formulation. Tiragolumab (formerly MTIG7192A) is a fully human IgG1 monoclonal antibiody derived in open monoclonal technology rats that binds to TIGIT and prevents its interaction with the poliovirus receptor. The recombinant antibody is produced in Chinese hamster ovary (CHO) cells and consists of two heavy chains (456 amino acid residues each) and two light chains (220 amino acid residues each).
32. Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment or within 6 months after the final dose of study treatment. Women of childbearing potential must have a negative serum pregnancy test result within 14 days prior to initiation of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-07-28 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
Safety and adverse events (AEs). | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Jianjun Zhang, MD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org